CLINICAL TRIAL: NCT03670329
Title: Efficacy and Acceptability of URGO2875 Dressing in the Treatment of Leg Ulcers With Inflammatory Signs
Brief Title: Management of Infection Risk in Non-comparative Trial (MINT)
Acronym: MINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-08-07-AWC008
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: Non-comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- URGO2875 (Experimental): Dressing
  Interventions: Device: URGO2875

INTERVENTIONS:
Device: URGO2875 — Dressing

SUMMARY:
The URGO2875 dressing is an innovative antimicrobial dressing made of exclusive technologies of TLC-Ag healing matrix and fibres. The dressing has been developed for the local treatment of chronic (leg ulcers, pressure ulcers, diabetic foot ulcers) and acute (burns, traumatic wounds, surgical wounds) moderately to highly exudative wounds at risk or with signs of local infection.

The purpose of this non-comparative clinical trial was to evaluate the performance (efficacy and safety) of the URGO2875 dressing, on the healing process of chronic wounds presenting a high-risk of infection.

DETAILED DESCRIPTION:
The URGO2875 dressing is indicated for the local treatment of chronic (leg ulcers, pressure ulcers, diabetic foot ulcers) and acute (burns, traumatic wounds, surgical wounds) moderately to highly exudative wounds at risk or with signs of local infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, aged ≥ 18 years, who signed and dated informed consent form,
* Patients affected by VLU or mixed ulcer of predominantly venous origin (ankle brachial pressure index (ABPI) ≥ 0.7 and ≤ 1.3),
* Patient willing and able to wear an effective venous compression system every day during the study period,
* Patient with at least three of the five inflammatory clinical signs : pain between dressing changes, periwound erythema, local oedema, malodour and presence of heavy exudate.

Exclusion Criteria:

* Patients under guardianship or protection of vulnerable adult
* Pregnancy or breastfeeding women,
* Childbearing potential women with no medically-acceptable method of birth control,
* Patients included in another clinical study,
* Patients with known allergy with hydrocolloid (carboxymethylcellulose CMC), silicone or silver,
* Patients with wound covered partially or totally with necrotic tissue,
* Patients who had within the 3 months prior the inclusion, deep vein thrombosis
* Patients with a serious general disease that deemed to interfere with the treatment period and evaluation
* Patients with progressive neoplastic lesions treated by radiotherapy, chemotherapy or hormone therapy
* Patients with non-controlled systemic infection by an suitable antibiotic therapy
* Patients with clinically infected wound
* Patients with wound requiring surgical treatment or for which surgery is scheduled during the study period
* Patients with known cancerous lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Wound surface area | 4 weeks
  Relative wound surface area reduction (%) at the end of the four weeks of treatment

SECONDARY OUTCOMES:
Inflammatory clinical signs | 4 weeks
  The decrease of the clinical score, based on the presence of the five inflammatory clinical signs,
Percentage of wounds with a favourable outcome | 4 weeks
  Defined as a relative wound area reduction of at least 40% after the 4-week treatment period
Time to healing | 4 weeks
  Wound Healing time in days
Healing | 4 weeks
  Percentage of Healing wound
Patient quality of life | 4 weeks
  Patient quality of life assessed with EuroQoL 5D-5L

OTHER OUTCOMES:
Adverse event | 4 weeks
  Adverse event related to the use of the testing dressing (serious/ non-serious) will be described.

CONTACTS AND LOCATIONS:
Overall Officials: GERI Ms Chloe, MD, Principal Investigator — Lapeyronie Hospital, Montpellier- FRANCE

IPD SHARING:
Plan to Share IPD: No